CLINICAL TRIAL: NCT00953628
Title: Endometrial Advancement After Rec or u-HCG Triggering
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Principal Investigator, Papanikolaou Evangelos, Lecturer Aristotle University Greece, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: recHCG001
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: endometrium; histology; pregnancy
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- o Group A=uHCG ovul trig (Active Comparator): HCG for triggering
  Interventions: Drug: 10000 IU urinary HCG
- o Group B=recHCG ovul trig (Experimental): recombinant HCG for triggering
  Interventions: Drug: 250 mcg recombinant HCG

INTERVENTIONS:
Drug: 10000 IU urinary HCG — bolus 10000 units for ovulation triggering
  Other Names: Pregnyl
  Arms: o Group A=uHCG ovul trig
Drug: 250 mcg recombinant HCG — bolus 250 mcg for ovulation triggering in IVF patients
  Other Names: Ovitrelle
  Arms: o Group B=recHCG ovul trig

SUMMARY:
The purpose of this study is to investigate any potential advantages of replacing human chorionic gonadotropin (uhCG) with recombinant human chorionic gonadotropin (recHCG) for final oocyte maturation with regard to Ovarian hyperstimulation syndrome (OHSS)pathophysiology, endometrium receptivity and embryo quality and clinical pregnancy.

DETAILED DESCRIPTION:
Biopsies of endometrium were taken in different groups Pregnancy rates were compared among defferent groups

ELIGIBILITY:
Inclusion Criteria:

* Less than 36 years old
* Male or tubal infertility
* FSH<12 on day 3

Exclusion Criteria:

* Endometriosis stage 3 & 4

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2005-08; Primary Completion 2006-12 (Actual); Study Completion 2008-12

PRIMARY OUTCOMES:
endometrium histology on the day of OPU | day of oocytre pick up

SECONDARY OUTCOMES:
pregnancy rate | 14 days after oocyte pick up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Devroey, Professor, Study Director — Professor or OB-GYN
Locations (1):
- Centre for Reproductive Medicine, UZ Brussel, Brussels, Jette, Belgium